CLINICAL TRIAL: NCT01647152
Title: A Pilot Study to Investigate Ustekinumab (StelaraTM) for the Treatment of Active Sight-Threatening Uveitis
Brief Title: Ustekinumab for Active Sight-Threatening Uveitis
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: National Eye Institute (NEI) (NIH)
Responsible Party: Sponsor
Organization: National Institutes of Health Clinical Center (CC) (NIH)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 120168; 12-EI-0168
Record Dates: First submitted 2012-07-19; First posted 2012-07-20 (Estimated); Last update posted 2019-12-05 (Actual); Status verified 2014-09-05

CONDITIONS: Uveitis
Keywords: Uveitis; Ustekinumab; IL 12/23; Stelara
MeSH Terms: conditions — Uveitis | interventions — Ustekinumab

INTERVENTIONS:
Drug: Ustekinumab

SUMMARY:
Background:

- Uveitis is an eye inflammation that can cause vision loss. It is treated with eye drops, drugs and sometimes surgery. In some people, treatment may not prevent vision loss. A type of white blood cells called T-cells often have a role in causing uveitis. In some cases of uveitis, T-cells attack the eye and cause inflammation. A drug called ustekinumab reduces inflammation from these T-cells. Researchers want to see if ustekinumab can be used to treat uveitis.

Objectives:

- To see if ustekinumab can be used to treat uveitis.

Eligibility:

- Individuals at least 18 years of age who have active uveitis that needs treatment.

Design:

* Participants will be screened with a physical exam, eye exam, and medical history. Blood and urine samples will be taken.
* Participants will have at least eight clinic visits during the 64-week study period. After the first visit, visits will occur at 2, 4, and 8 weeks, and then every 12 weeks.
* Participants will have a ustekinumab injection at the first study visit. They will have additional doses at the second and third visits, and then every 12 weeks until 1 year after the first dose (Week 52).
* Treatment will be monitored with frequent blood tests and eye exams. Other standard treatments for uveitis may be given as needed.
* There will be a final study visit 3 months after the last injection.

DETAILED DESCRIPTION:
Objective: Uveitis refers to intraocular inflammatory diseases that are an important cause of visual loss. Standard systemic immunosuppressive medications for uveitis can cause significant adverse effects and many patients continue to experience disease flare-ups. Ustekinumab is a human IL-12 and -23 antagonist. The involvement of IL-12 and IL-23 in the pathophysiology of uveitis and other autoimmune diseases known to be associated with uveitis suggests that ustekinumab could be a potential treatment for uveitis. The study objective is to investigate the safety, tolerability and potential efficacy of subcutaneous injections of ustekinumab as a possible treatment for active intermediate uveitis, posterior uveitis or panuveitis.

Study Population: Five participants with active intermediate uveitis, posterior uveitis or panuveitis who meet the inclusion criteria will be initially enrolled. Up to seven participants may be enrolled, as up to two participants may be accrued to account for participants who withdraw from the study prior to Week 8.

Design: This is a prospective, non-randomized, uncontrolled, single-center pilot study to evaluate subcutaneous injections of ustekinumab as a possible treatment for active intermediate uveitis, posterior uveitis or panuveitis. Participants will receive a 90 mg subcutaneous injection of ustekinumab at baseline and a second and third injection at Week 2 and 4 and every 12 weeks thereafter. Participants will continue to receive injections of ustekinumab every 12 weeks until Week 52. Participants will return for a final safety visit 12 weeks later.

Outcome Measures: The primary outcome is the number of participants who experience treatment response (as defined in Appendix 1) by Week 8. Secondary outcomes include changes in visual acuity, the number of participants who experience a recurrence, the number of days to recurrence, presence or extent of macular edema, the amount of retino-vascular leakage, changes in retinal thickening, the length of time to quiescence and the ability to taper concomitant immunosuppressive medications. Safety outcomes include the number and severity of systemic and ocular toxicities and adverse events, the proportion of participants who experience vision loss of greater than or equal to 15 Early Treatment Diabetic Retinopathy Study (ETDRS) letters and the number of participants who experience a substantial rise in elevated intraocular pressure (IOP).

ELIGIBILITY:
* INCLUSION CRITERIA:

  1. Participant has the ability to understand and sign the informed consent document.
  2. Participant is 18 years of age or older.
  3. Participant has negative PPD or quantiferon testing done within three months prior to enrollment or had latent TB but has completed prophylactic anti-TB treatment.
  4. Participant has active intermediate uveitis, posterior uveitis or panuveitis in at least one eye requiring systemic therapy. Active disease is defined as:

     * 1 or more anterior chamber cells (according to SUN criteria); and/or
     * 0.5 or more vitreous haze (according to SUN criteria); and/or

     Active chorioretinitis or greater than or equal to quadrants with leakage on FA.
  5. Participant has visual acuity in at least one eye of 20/400 or better.
  6. Participant is willing and able to comply with the study procedures.
  7. Female participants of childbearing potential must not be pregnant or breast-feeding, have a negative pregnancy test at screening and must be willing to undergo pregnancy testing throughout the study.
  8. Both female participants of childbearing potential and male participants able to father a child must have (or have a partner who has) had a hysterectomy or vasectomy, be completely abstinent from intercourse or must agree to practice two effective methods of contraception throughout the course of the study and for six weeks after the last investigational product injection. Acceptable methods of contraception for this study include:
* hormonal contraception (i.e., birth control pills, injected hormones, dermal patch or vaginal ring),
* intrauterine device,
* barrier methods (diaphragm, condom) with spermicide, or
* surgical sterilization (tubal ligation).

EXCLUSION CRITERIA:

1. Participant has a significant active infection (an infection requiring treatment as determined by the medical team), including active tuberculosis or human immunodeficiency virus (HIV).
2. Participant received a live vaccination within the past six weeks.
3. Participant is expected to receive a live vaccination at any time during the study.
4. Participant received the Bacillus Calmette-Guerin (BCG) vaccine within the past year.
5. Participant is expected to receive the BCG vaccine at anytime during the study or up to one year after discontinuing ustekinumab.
6. Participant has a history of cancer (other than a non-melanoma skin cancer) diagnosed within the past five years.
7. Participant has received intraocular (or periocular) steroid or anti-VEGF injections within the last six weeks.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2012-07-03; Primary Completion 2015-06-30 (Estimated); Study Completion 2015-06-30 (Estimated)

PRIMARY OUTCOMES:
The primary outcome is the number of participants who experience at least a 2-step (or down to grade 0) reduction in inflammation as per the Standardization of Uveitis Nomenclature (SUN) criteria by Week 8.

CONTACTS AND LOCATIONS:
Overall Officials: Hatice N Sen, M.D., Principal Investigator — National Eye Institute (NEI)

REFERENCES:
- [Background] Gritz DC, Wong IG. Incidence and prevalence of uveitis in Northern California; the Northern California Epidemiology of Uveitis Study. Ophthalmology. 2004 Mar;111(3):491-500; discussion 500. doi: 10.1016/j.ophtha.2003.06.014. PMID 15019324
- [Background] Djalilian AR, Nussenblatt RB. Immunosuppression in uveitis. Ophthalmol Clin North Am. 2002 Sep;15(3):395-404, viii. doi: 10.1016/s0896-1549(02)00036-6. PMID 12434489
- [Background] Luger D, Silver PB, Tang J, Cua D, Chen Z, Iwakura Y, Bowman EP, Sgambellone NM, Chan CC, Caspi RR. Either a Th17 or a Th1 effector response can drive autoimmunity: conditions of disease induction affect dominant effector category. J Exp Med. 2008 Apr 14;205(4):799-810. doi: 10.1084/jem.20071258. Epub 2008 Apr 7. PMID 18391061